CLINICAL TRIAL: NCT04397445
Title: Clinical Study to Investigate the Urinary Excretion of N-nitrosodimethylamine (NDMA) After Ranitidine Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SCR-010
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Ranitidine Adverse Reaction; Pharmacokinetics; Food-drug Interaction
Keywords: Ranitidine; N-nitrosodimethylamine; NDMA; Urine excretion
MeSH Terms: interventions — Ranitidine

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, single-dose, 4-period crossover study with 18 healthy subjects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing. Subjects and staff will be blinded to treatment assignment. The blind will be maintained through a randomization schedule held by the dispensing pharmacist. Subjects will be blindfolded during oral study drug administration. All subjects will be provided low nitrite/NDMA meals for the first two periods of the study and high nitrite/NDMA meals for the last two periods of the study. This ordering of meals will allow purchasing a single lot of perishable items for different meals and to simplify meal preparation and serving at the study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ranitidine and Low Nitrite/NDMA Meals (Noncured-Meats Diet) (Experimental): Single dose of ranitidine (300 mg) plus low nitrite/NDMA meals (noncured-meats diet)
  Interventions: Drug: Ranitidine; Other: Low nitrite/NDMA meals
- Placebo and Low Nitrite/NDMA Meals (Noncured-Meats Diet) (Placebo Comparator): Single dose of placebo plus low nitrite/NDMA meals (noncured-meats diet)
  Interventions: Drug: Placebo; Other: Low nitrite/NDMA meals
- Ranitidine and High Nitrite/NDMA Meals (Cured-Meats Diet) (Experimental): Single dose of ranitidine (300 mg) plus high nitrite/NDMA meals (cured-meats diet)
  Interventions: Drug: Ranitidine; Other: High nitrite/NDMA meals
- Placebo and High Nitrite/NDMA Meals (Cured-Meats Diet) (Placebo Comparator): Single dose of placebo plus high nitrite/NDMA meals (cured-meats diet)
  Interventions: Drug: Placebo; Other: High nitrite/NDMA meals

INTERVENTIONS:
Drug: Ranitidine — Ranitidine 300 mg
  Arms: Ranitidine and High Nitrite/NDMA Meals (Cured-Meats Diet); Ranitidine and Low Nitrite/NDMA Meals (Noncured-Meats Diet)
Drug: Placebo — Oral placebo tablet
  Arms: Placebo and High Nitrite/NDMA Meals (Cured-Meats Diet); Placebo and Low Nitrite/NDMA Meals (Noncured-Meats Diet)
Other: Low nitrite/NDMA meals — Meals containing low levels of nitrites and NDMA
  Other Names: Noncured-meats diet
  Arms: Placebo and Low Nitrite/NDMA Meals (Noncured-Meats Diet); Ranitidine and Low Nitrite/NDMA Meals (Noncured-Meats Diet)
Other: High nitrite/NDMA meals — Meals containing higher levels of nitrites and NDMA
  Other Names: Cured-meats diet
  Arms: Placebo and High Nitrite/NDMA Meals (Cured-Meats Diet); Ranitidine and High Nitrite/NDMA Meals (Cured-Meats Diet)

SUMMARY:
Ranitidine is an over-the-counter and prescription drug, which decreases the amount of acid secreted by the stomach. Some ranitidine medicines contain an impurity called N-nitrosodimethylamine (NDMA) at low levels. NDMA is classified as a probable human carcinogen (a substance that could cause cancer) based on results from laboratory tests. NDMA is a known environmental contaminant and found in water and foods, including meats, dairy products, and vegetables.

The US Food and Drug Administration (FDA) has found levels of NDMA in some ranitidine products similar to the levels you would expect to be exposed to if you ate common foods like grilled or smoked meats. The ranitidine that will be used in this study has been tested twice (months apart) and shown to have stable NDMA levels well below the acceptable daily limit. Of note, the risk of NDMA with ranitidine is only relevant with prolonged chronic administration as at the acceptable limit, there is approximately a 1 in 100,000 chance of cancer after 70 years of exposure to that level.

FDA has also conducted tests that simulate the potential formation of NDMA from ranitidine after it has been exposed to acid in the stomach with a normal diet. Results of these tests indicate that NDMA is not formed in typical stomach conditions. Similarly, if ranitidine is exposed to a simulated small intestinal fluid, NDMA is not formed. Other laboratory experiments suggest a combination of nitrites, such as found in processed meats, and an acidic environment may increase NDMA formation, however the levels of nitrites tested were very high. Separately, a previous study in 10 healthy volunteers showed that volunteers who received ranitidine had an increase in urinary NDMA excreted over 24 h. The level of increase was greater than would be expected from laboratory testing.

This clinical study is being performed to determine if and how much NDMA is produced from ranitidine in the human body and whether nitrite-containing foods may increase formation of NDMA. The study will use a prescription dose of ranitidine (300 mg) to test whether there is increased urinary NDMA excretion levels over 24-hours after ranitidine administration in comparison to placebo when participants are administered low nitrite/NDMA meals and when subjects are administered high nitrite/NDMA meals. On 4 different days, each participant will receive ranitidine or placebo with high nitrite/NDMA meals and ranitidine or placebo with low nitrite/NDMA meals.

DETAILED DESCRIPTION:
The U.S. Food and Drug Administration (FDA) has learned that some ranitidine medicines, including some products commonly known as the brand-name drug Zantac, contain a nitrosamine impurity called N-nitrosodimethylamine (NDMA) at low levels. NDMA is classified as a probable human carcinogen (a substance that could cause cancer) based on results from laboratory tests. NDMA is a known environmental contaminant and found in water and foods, including meats, dairy products, and vegetables.

The FDA has been investigating NDMA and other nitrosamine impurities in blood pressure and heart failure medicines called Angiotensin II Receptor Blockers (ARBs) since 2018. In the case of ARBs, the FDA has recommended numerous recalls as it discovered unacceptable levels of nitrosamines.

FDA has found levels of NDMA in ranitidine active pharmaceutical ingredient and finished drugs that are similar to the levels you would expect to be exposed to if you ate common foods like grilled or smoked meats. FDA has requested removal of all ranitidine products from the market because some ranitidine products have NDMA levels above the acceptable limits (96 nanograms per day or 0.32 parts per million for 300 mg per day of ranitidine) and that levels of NDMA in ranitidine may increase to unacceptable levels over time. However, FDA has not withdrawn approvals of ranitidine new drug applications and abbreviated new drug applications and if a company can show, through scientific data, that their ranitidine product is stable and the NDMA levels do not increase over time to unsafe levels, FDA may consider allowing that ranitidine product back on the U.S. market. The ranitidine that will be used in this study has been tested twice (months apart) and shown to have stable NDMA levels well below the acceptable daily limit. Of note, the risk of NDMA with ranitidine is only relevant with prolonged chronic administration as at the acceptable limit, there is approximately a 1 in 100,000 chance of cancer after 70 years of exposure to that level.

FDA has also conducted tests that simulate the potential formation of NDMA from ranitidine after it has been exposed to acid in the stomach with a normal diet. Results of these tests indicate that NDMA is not formed in typical stomach conditions. Similarly, if ranitidine is exposed to a simulated small intestinal fluid, NDMA is not formed. Other in vitro experiments suggest a combination of nitrites, such as found in processed meats, and an acidic environment potentiate formation of NDMA. For that reason, prior to requesting removal of ranitidine products from the market, the FDA had advised consumers who wished to continue taking these medications to consider limiting consumption of nitrite-containing foods.

Separately, a previous study in 10 healthy volunteers showed that single dose administration of ranitidine 150 mg was associated with ~400-fold increase in urinary NDMA excreted over 24 h. This level of increase is substantially greater than would be expected from laboratory testing. Further evaluation is necessary to determine if and how much NDMA is produced from ranitidine in the human body and whether nitrite-containing foods may potentiate formation of NDMA in vivo.

Ranitidine

Ranitidine is an over-the-counter (OTC) and prescription drug. Ranitidine is an histamine-2 (H2) blocker, which decreases the amount of acid secreted by the stomach. Over-the-counter ranitidine is approved to prevent and relieve heartburn associated with acid ingestion and sour stomach and the approved dosage regiment is up to 150 mg twice a day. Prescription ranitidine is approved for multiple indications, including treatment and prevention of ulcers of the stomach and intestines and treatment of gastroesophageal reflux disease and the approved dosage regimen is up to 150 mg twice a day or 300 mg once a day.

Study Primary Objective

1. To evaluate 24-hour urinary excretion of NDMA after oral administration of ranitidine compared to placebo

Study Exploratory Objectives

1. To evaluate plasma ranitidine, NDMA, and dimethylamine (DMA) after oral administration of ranitidine compared to placebo
2. To evaluate urinary excretion amounts over 24-hours of ranitidine and DMA after oral administration of ranitidine compared to placebo
3. To evaluate 24-hour urinary excretion and plasma concentration of NDMA and DMA with administration of high nitrite/NDMA meals compared to low nitrite/NDMA meals

Study Design

This is a randomized, placebo-controlled, single-dose, 4-period crossover study with 18 healthy subjects. Subjects check-in on Day -2 and receive the following 4 treatments starting on Day 1, with one washout day between treatment days. The treatments consist of oral administration of either a single dose of ranitidine (300 mg) or placebo administered at time 0 hr. All subjects will be provided low nitrite/NDMA meals for the first two periods of the study and high nitrite/NDMA meals for the last two periods of the study. This ordering of meals will allow purchasing a single lot of perishable items for different meals and to simplify meal preparation and serving at the study site. The four treatments are:

A. Ranitidine + low nitrite/NDMA meal;

B. Placebo + low nitrite/NDMA meal;

C. Ranitidine + high nitrite/NDMA meal;

D. Placebo + high nitrite/NDMA meal.

Subjects will report to the study site for screening from Days -28 to -3 and then will return to the site on Day -2 for baseline assessments. Subjects will receive three standardized meals and an evening snack per day starting on Day -1. Subjects will be served meals from a pre-specified menu for check-in and for all washout and treatment days. Subjects will be instructed to finish all their meals within 25 minutes with no leftovers. Subjects will only consume foods served to them at planned meal and snack times.

Two different full day menus of low nitrite/NDMA and high nitrite/NDMA meals have been developed. Additional details regarding the meals will be specified in the Meal Preparation Plan. Meals will be identical for treatments A and B (low nitrite/NDMA meal) of the study and a separate set of identical low nitrite/NDMA meals will be served on the washout days prior to treatment. Likewise, meals will be identical for treatments C and D (high nitrite/NDMA meal) and a separate set of identical high nitrite/NDMA meals will be served on the washout days prior to treatment. The last meal on Day -1, Day 2, Day 4, and Day 6 should be administered at approximately 18:00 to permit at least 12-hour fasting prior to dosing. Outside of meal times, subjects will be provided with distilled water to drink throughout the study.

On study treatment days, the first meal will be provided at the time of dosing. Subjects will be instructed to swallow the medication with approximately 250 mL of room temperature distilled water and begin eating one minute after dosing. Subjects are required to eat each meal in its entirety during the study. If the meal is not finished, the reason should be recorded, along with what was not eaten, and a picture of the remaining food should be taken.

Prior to and following study drug or placebo administration on Day 1, subjects will undergo assessments as described in the Schedule of Events. There will be one day of washout between periods. Participants will be confined in the study clinic from Day -2 until the morning of Day 8.

During the screening visit, the inclusion and exclusion criteria will be reviewed to ensure the subject is eligible for the study. Subjects will be shown the low and high nitrite/NDMA menus and informed that each meal in the menu must be finished in its entirety. The subject must agree to consume all planned meals in order to be eligible to participate. The informed consent form will be reviewed with the subject by a member of the study team and the subject will be encouraged to ask questions to ensure he or she has a good understanding of the study. If the subject is eligible and agrees to participate, the subject will be asked to sign the informed consent form before any study specific procedure is performed, including randomization. Results of all screening tests will be evaluated by the study clinician/investigator against the inclusion/exclusion criteria to confirm subject eligibility. For subjects that are eligible, a molecular diagnostic test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) will be performed just before or at check-in.

During the study, urine and blood samples for pharmacokinetic assessments will occur before or after drug or placebo administration at the following timepoints:

* Urine samples will be collected using separate collection containers over 24 h. Collection times will occur at 0 (pre-dose), 3, 6, 9, 12, 15, and 24 h. Subjects will be instructed to void their bladder at each collection time and total weight of the sample will be recorded. If a subject must void their bladder at an unscheduled time, the unscheduled voids will be collected, and total weight of the unscheduled voiding will be recorded. The unscheduled voiding sample will be treated, analytically analyzed, and reported as part of scheduled sample collection for determining cumulative amounts of NDMA, ranitidine, and DMA excreted over 24 h.
* Plasma samples will be collected at 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 11, 14, and 24 h post-dose.

Subjects will be discharged from the study after completion of all study procedures. If a subject discontinues from the study prematurely, all procedures scheduled for the end of the study will be performed. Meals (timing and components), activity levels, and general conditions in the study clinic will be standardized to the extent possible on the treatment days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to sign an institutional review board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy, non-smoking man or woman, 18 to 50 years of age, inclusive, who has a body mass index (BMI) of 18.5 to 32 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and Check-in (Day -2).
5. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day -2) and agree to remain strictly abstinent for the duration of the study and for at least 1 month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -2) until at least 1 month after the end of the study.
6. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Subject has used antacids or proton pump inhibitors within 14 days of screening (interferes with H. pylori testing).
2. Subject has used any prescription or nonprescription drugs (including antacids, proton pump inhibitors, aspirin or non-steroidal anti-inflammatory drugs [NSAIDs] and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug.
3. Subject is currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
4. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening.
5. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, cola), caffeine, grapefruit, or grapefruit juice within 24 h of check-in. Subjects must refrain from ingesting these throughout the study. Subjects must also refrain from using mouthwash from check-in until check-out.
6. Subject has a history or evidence of a clinically significant disorder, condition, or disease (e.g., cancer, human immunodeficiency virus [HIV], hepatic or renal impairment) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion. This includes subjects with any underlying medical conditions that put subjects at higher risk for coronavirus disease of 2019 (COVID-19) complications; per current Center for Disease Control and Prevention (CDC) recommendations this includes:

   * People with chronic lung disease or moderate to severe asthma
   * People who have serious heart conditions
   * People who are immunocompromised
   * Many conditions can cause a person to be immunocompromised, including cancer treatment, smoking, bone marrow or organ transplantation, immune deficiencies, poorly controlled HIV, and prolonged use of corticosteroids and other immune weakening medications
   * People with severe obesity (BMI of 40 kg/m2 or higher)
   * People with diabetes
   * People with chronic kidney disease undergoing dialysis
   * People with liver disease
7. Subject has any signs or symptoms that are consistent with COVID-19. Per current CDC recommendations this includes subjects with the symptoms cough or shortness of breath or difficulty breathing, or at least two of the following symptoms: fever, chills, repeated shaking with chills, muscle pain, headache, sore throat or new loss of taste/smell. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
8. Subject tests positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by a molecular diagnostic test performed prior to admission.
9. Subject has known or suspected allergies or sensitivities to the study drug.
10. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at Screening or Check-In that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
11. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
12. Subject has a history of H. pylori infection or ulcer disease or has a positive breath test for H. pylori at screening.
13. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
14. Female subjects are pregnant or lactating before enrollment in the study.
15. Subject is not willing to eat all of every meal that will be served during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Nalepinski, MPAS, PA-C, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as part of a manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as with any eventual publications.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Florian J, Matta MK, DePalma R, Gershuny V, Patel V, Hsiao CH, Zusterzeel R, Rouse R, Prentice K, Nalepinski CG, Kim I, Yi S, Zhao L, Yoon M, Selaya S, Keire D, Korvick J, Strauss DG. Effect of Oral Ranitidine on Urinary Excretion of N-Nitrosodimethylamine (NDMA): A Randomized Clinical Trial. JAMA. 2021 Jul 20;326(3):240-249. doi: 10.1001/jama.2021.9199. PMID 34180947
- See also: FDA Updates and Press Announcements on NDMA in Zantac (ranitidine). — https://www.fda.gov/drugs/drug-safety-and-availability/fda-updates-and-press-announcements-ndma-zantac-ranitidine
- See also: Ranitidine Package Insert updated December 7, 2018. — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=4654adbd-c107-4846-9ee6-13f314bc2798
- See also: Zeng T, Mitch WA. Oral intake of ranitidine increases urinary excretion of N-nitrosodimethylamine. Carcinogenesis. 2016 Jun;37(6):625-634. doi: 10.1093/carcin/bgw034. Epub 2016 Mar 18. — https://pubmed.ncbi.nlm.nih.gov/26992900/

RESULTS

PARTICIPANT FLOW:
Groups:
- ABCD: Participants first received a single dose of ranitidine, 300 mg, with a noncured meats diet designed to contain lower amounts of nitrites, nitrates (nitrate-reducing bacteria can convert nitrates to nitrites), and NDMA (Treatment A), then crossed over to the sequential treatments with one day of washout in between treatments.
  Treatment B: Single dose of oral placebo with a noncured meats diet designed to contain lower amounts of nitrites, nitrates, and NDMA
  Treatment C: Single dose of ranitidine, 300 mg with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
  Treatment D: Single dose of oral placebo with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
- BACD: Participants first received a single dose of oral placebo with a noncured meats diet designed to contain lower amounts of nitrites, nitrates (nitrate-reducing bacteria can convert nitrates to nitrites), and NDMA (Treatment B), then crossed over to the sequential treatments with one day of washout in between treatments.
  Treatment A: Single dose of oral ranitidine, 300 mg, with a noncured meats diet designed to contain lower amounts of nitrites, nitrates, and NDMA
  Treatment C: Single dose of ranitidine, 300 mg with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
  Treatment D: Single dose of oral placebo with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
- ABDC: Participants first received a single dose of ranitidine, 300 mg, with a noncured meats diet designed to contain lower amounts of nitrites, nitrates (nitrate-reducing bacteria can convert nitrates to nitrites), and NDMA (Treatment A), then crossed over to the sequential treatments with one day of washout in between treatments.
  Treatment B: Single dose of oral placebo with a noncured meats diet designed to contain lower amounts of nitrites, nitrates, and NDMA
  Treatment D: Single dose of oral placebo with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
  Treatment C: Single dose of ranitidine, 300 mg with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
- BADC: Participants first received a single dose of oral placebo with a noncured meats diet designed to contain lower amounts of nitrites, nitrates (nitrate-reducing bacteria can convert nitrates to nitrites), and NDMA (Treatment B), then crossed over to the sequential treatments with one day of washout in between treatments.
  Treatment A: Single dose of oral ranitidine, 300 mg, with a noncured meats diet designed to contain lower amounts of nitrites, nitrates, and NDMA
  Treatment D: Single dose of oral placebo with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
  Treatment C: Single dose of ranitidine, 300 mg with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
Period: Overall Study
Arm/Group | ABCD | BACD | ABDC | BADC
Started | 5 | 5 | 4 | 4
Completed | 4 | 5 | 4 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were randomized to 1 of 4 treatment sequences (i.e., ABCD, BACD, ABDC, and BADC) and over 4 periods received ranitidine (300 mg) and placebo (randomized order) with a noncured-meats diet and then a cured-meats diet.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.0 [28.3 to 42.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Body Weight [Median (Inter-Quartile Range); unit: kg] | 76.9 [62.6 to 83.7]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative NDMA Amount Excreted in Urine Over 24 Hours After Drug Administration (Comparison Between Ranitidine and Placebo)
Description: The cumulative amount of NDMA excreted over 24 hours is determined by calculating the amount excreted during specified intervals (includes all planned collections and unscheduled voids) and summarizing totals over a 24-h period.
Time Frame: 24-hours post-dose including planned collections (at 3, 6, 9, 12, 15, and 24 hours post-dose) and unscheduled voids. All subjects voided at approximately 0 hours (pre-dose), which was not included in the assessment.
Population: All participants who completed two paired treatment periods (i.e., ranitidine and placebo with the same diet)
Measure: Median (Inter-Quartile Range); unit: nanograms
Groups:
- Ranitidine and Noncured Meats Diet: Single dose of ranitidine, 300 mg with a noncured meats diet designed to contain lower amounts of nitrites, nitrates, and NDMA
- Placebo and Noncured Meats Diet: Single dose of oral placebo with a noncured meats diet designed to contain lower amounts of nitrites, nitrates, and NDMA
- Ranitidine and Cured Meats Diet: Single dose of ranitidine, 300 mg with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
- Placebo and Cured Meats Diet: Single dose of oral placebo with a cured meats diet designed to contain higher amounts of nitrites, nitrates, and NDMA
Arm/Group | Ranitidine and Noncured Meats Diet | Placebo and Noncured Meats Diet | Ranitidine and Cured Meats Diet | Placebo and Cured Meats Diet
Number analyzed (Participants) | 17 | 17 | 17 | 17
nanograms | 0.6 [0 to 29.7] | 10.5 [0 to 17.8] | 11.9 [5.6 to 48.6] | 23.4 [8.6 to 36.7]
Statistical Analysis 1: Comparison: Ranitidine and Noncured Meats Diet vs Placebo and Noncured Meats Diet; A Wilcoxon signed-rank test was used for analyses, per the statistical analysis plan, as NDMA urine data were not normally distributed; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney) — A 1-sided lower P value <.05 was considered significant for ranitidine vs. placebo as the aim was to evaluate if ranitidine increased NDMA exposure. Comparisons were performed separately with each diet without adjustment for multiplicity; The median of the paired differences (interquartile range) between ranitidine and placebo is 0 (-6.9 to 0) ng. The median of the paired differences is calculated by first determining the difference between the two treatments for each individual participant and then determining the median of those values. The Wilcoxon signed-rank test that was used for NDMA analyses is also based on first determining the difference between the treatment groups for each individual participant
Statistical Analysis 2: Comparison: Ranitidine and Cured Meats Diet vs Placebo and Cured Meats Diet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; The median of the paired differences (interquartile range) between ranitidine and placebo is -1.1 (-9.1 to 11.5) ng. The median of the paired differences is calculated by first determining the difference between the two treatments for each individual participant and then determining the median of those values. The Wilcoxon signed-rank test that was used for NDMA analyses is also based on first determining the difference between the treatment groups for each individual participant

2. Other Pre Specified Outcome: Cumulative NDMA Amount Excreted in Urine Over 24 Hours After Drug Administration (Comparison Between Diets)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All participants who completed two paired treatment periods (i.e., ranitidine and placebo with the same diet)
Measure: Median (Inter-Quartile Range); unit: nanograms
Arm/Group | Ranitidine and Cured Meats Diet | Ranitidine and Noncured Meats Diet | Placebo and Cured Meats Diet | Placebo and Noncured Meats Diet
Number analyzed (Participants) | 17 | 17 | 17 | 17
nanograms | 11.9 [5.6 to 48.6] | 0.6 [0 to 29.7] | 23.4 [8.6 to 36.7] | 10.5 [0 to 17.8]
Statistical Analysis 1: Comparison: Ranitidine and Cured Meats Diet vs Ranitidine and Noncured Meats Diet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney) — Exploratory analyses on the effect of diet used a 1-sided lower P value <.05 for NDMA as the cured-meats diet was designed to have higher NDMA; The median of the paired differences (interquartile range) between the cured-meats diet and noncured-meats diet is 9.3 (3.8 to 25.0) ng. The median of the paired differences is calculated by first determining the difference between the two treatments for each individual participant and then determining the median of those values. The Wilcoxon signed-rank test that was used for NDMA analyses is also based on first determining the difference between the treatment groups for each individual participant
Statistical Analysis 2: Comparison: Placebo and Cured Meats Diet vs Placebo and Noncured Meats Diet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; The median of the paired differences (interquartile range) between the cured-meats diet and noncured-meats diet is 6.4 (0 to 23.4) ng. The median of the paired differences is calculated by first determining the difference between the two treatments for each individual participant and then determining the median of those values. The Wilcoxon signed-rank test that was used for NDMA analyses is also based on first determining the difference between the treatment groups for each individual participant

3. Other Pre Specified Outcome: Cumulative Dimethylamine (DMA) Amount Excreted in Urine Over 24 Hours After Drug Administration
Description: The cumulative amount of DMA excreted over 24 hours is determined by calculating the amount excreted during specified intervals (includes all planned collections and unscheduled voids) and summarizing totals over a 24-h period.
Time Frame: as for outcome 1
Population: All participants who completed two paired treatment periods (i.e., ranitidine and placebo with the same diet)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Ranitidine and Noncured Meats Diet | Placebo and Noncured Meats Diet | Ranitidine and Cured Meats Diet | Placebo and Cured Meats Diet
Number analyzed (Participants) | 17 | 17 | 17 | 17
milligrams | 38.8 (38) | 41.1 (33) | 40.7 (52) | 43.1 (34)
Statistical Analysis 1: Comparison: Ranitidine and Noncured Meats Diet vs Placebo and Noncured Meats Diet; As DMA data were log-normally distributed, analyses were based on a mixed-effect analysis of geometric means with terms for treatment, period, and sequence; Test type: Other; p = 0.92, Mixed Models Analysis — A 1-sided lower P value <.05 was considered significant for the exploratory analyses of ranitidine vs. placebo because the study aim was to evaluate if ranitidine increased DMA exposure; Geometric Mean Ratio = 0.94, 90% CI 2-sided [0.87 to 1.01] — This compares the results from ranitidine (numerator) with placebo (denominator)
Statistical Analysis 2: Comparison: Ranitidine and Cured Meats Diet vs Placebo and Cured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.74, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 0.95, 90% CI 2-sided [0.81 to 1.10] — This compares the results from ranitidine (numerator) with placebo (denominator)
Statistical Analysis 3: Comparison: Ranitidine and Noncured Meats Diet vs Ranitidine and Cured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.52, Mixed Models Analysis — A 2-sided P value <.05 was used for DMA as the diet was not expected to affect these outcomes; Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.90 to 1.23] — This compares the results from the cured-meats diet (numerator) with the noncured-meats diet (denominator)
Statistical Analysis 4: Comparison: Placebo and Noncured Meats Diet vs Placebo and Cured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.42, Mixed Models Analysis — A 2-sided P value <.05 was used for DMA as the diet was not expected to affect these outcomes; Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.93 to 1.19] — This compares the results from the cured-meats diet (numerator) with the noncured-meats diet (denominator)

4. Other Pre Specified Outcome: Cumulative Ranitidine Amount Excreted in Urine Over 24 Hours After Drug Administration
Description: The cumulative amount of ranitidine excreted over 24 hours is determined by calculating the amount excreted during specified intervals (includes all planned collections and unscheduled voids) and summarizing totals over a 24-h period.
Time Frame: as for outcome 1
Population: All participants who completed two paired treatment periods (i.e., ranitidine and placebo with the same diet)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Ranitidine and Cured Meats Diet | Ranitidine and Noncured Meats Diet
Number analyzed (Participants) | 17 | 17
milligrams | 91.7 (29) | 74.1 (39)
Statistical Analysis 1: Comparison: Ranitidine and Cured Meats Diet vs Ranitidine and Noncured Meats Diet; As ranitidine data were log-normally distributed, analyses were based on a mixed-effect analysis of geometric means with terms for treatment, period, and sequence; Test type: Other; p = 0.001, Mixed Models Analysis — Exploratory analyses on the effect of diet used a 2-sided P value <.05 for ranitidine as the diet was not expected to affect these outcomes; Geometric Mean Ratio = 0.81, 95% CI 2-sided [0.72 to 0.91]; This compares the results from the cured-meats diet (numerator) with the noncured-meats diet (denominator)

5. Other Pre Specified Outcome: Area Under the Curve From Time Zero to the Last Sample Time (AUC(0-t)) of Plasma NDMA
Description: Determined for each subject using non-compartmental methods. All parameters will be reported with standard descriptive statistics including the geometric mean and coefficient of variation. Calculation of pharmacokinetic parameters will be performed using actual sampling times over a 24-h period.
Time Frame: 24-hours post-dose with planned samples at 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 11, 14, and 24 h post-dose
Population: All participants who completed two paired treatment periods (i.e., ranitidine and placebo with the same diet) and with sufficient data for calculating pharmacokinetic parameters. Note: AUC could not be calculated for NDMA for any participant during any period. The majority of samples (87-91% of plasma samples by period) were below the lower limit of quantification. The NDMA plasma profiles did not show sustained quantifiable amounts of NDMA and thus did not support calculation of an AUC.
Arm/Group | Ranitidine and Noncured Meats Diet | Placebo and Noncured Meats Diet | Ranitidine and Cured Meats Diet | Placebo and Cured Meats Diet
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: AUC(0-t) of Plasma DMA
Description: as for outcome 5
Time Frame: 24-hours post-dose with planned samples at 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 11, 14, and 24 h post-dose
Population: All participants who completed two paired treatment periods (i.e., ranitidine and placebo with the same diet) and with sufficient data for calculating pharmacokinetic parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter
Arm/Group | Ranitidine and Noncured Meats Diet | Placebo and Noncured Meats Diet | Ranitidine and Cured Meats Diet | Placebo and Cured Meats Diet
Number analyzed (Participants) | 17 | 17 | 17 | 17
micrograms*hour/milliliter | 26.3 (34) | 26.2 (35) | 20.9 (53) | 20.9 (46)
Statistical Analysis 1: Comparison: Ranitidine and Noncured Meats Diet vs Placebo and Noncured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.46, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 1.00, 90% CI 2-sided [0.91 to 1.11] — This compares the results from ranitidine (numerator) with placebo (denominator)
Statistical Analysis 2: Comparison: Ranitidine and Cured Meats Diet vs Placebo and Cured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.49, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 1.00, 90% CI 2-sided [0.80 to 1.25]; This compares the results from ranitidine (numerator) with placebo (denominator)
Statistical Analysis 3: Comparison: Ranitidine and Noncured Meats Diet vs Ranitidine and Cured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.02, Mixed Models Analysis — A 2-sided P value <.05 was used for DMA as the diet was not expected to affect these outcomes; Geometric Mean Ratio = 0.80, 95% CI 2-sided [0.67 to 0.95] — This compares the results from the cured-meats diet (numerator) with the noncured-meats diet (denominator)
Statistical Analysis 4: Comparison: Placebo and Noncured Meats Diet vs Placebo and Cured Meats Diet; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.03, Mixed Models Analysis — A 2-sided P value <.05 was used for DMA as the diet was not expected to affect these outcomes; Geometric Mean Ratio = 0.80, 95% CI 2-sided [0.65 to 0.98]; This compares the results from the cured-meats diet (numerator) with the noncured-meats diet (denominator)

7. Other Pre Specified Outcome: AUC(0-t) of Plasma Ranitidine
Description: as for outcome 5
Time Frame: 24-hours post-dose with planned samples at 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 11, 14, and 24 h post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter
Arm/Group | Ranitidine and Cured Meats Diet | Ranitidine and Noncured Meats Diet
Number analyzed (Participants) | 17 | 17
nanograms*hour/milliliter | 3736 (29) | 4857 (21)
Statistical Analysis 1: Comparison: Ranitidine and Cured Meats Diet vs Ranitidine and Noncured Meats Diet; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.66 to 0.89] — This compares the results from the cured-meats diet (numerator) with the noncured-meats diet (denominator)

ADVERSE EVENTS:
Time Frame: 10 days
Groups:
- Lead-in (No Treatment): Participants checked in one day early in order to standardize meals given the day prior to treatment start.
- Ranitidine and Noncured Meats Diet: Single dose of ranitidine (300 mg) plus low nitrite/NDMA meals
  Ranitidine: Ranitidine 300 mg
  Low nitrite/NDMA meals: Meals containing low levels of nitrites and NDMA (noncured meats diet)
- Placebo and Noncured Meats Diet: Single dose of placebo plus low nitrite/NDMA meals
  Placebo: Oral placebo tablet
  Low nitrite/NDMA meals: Meals containing low levels of nitrites and NDMA (noncured meats diet)
- Ranitidine and Cured Meats Diet: Single dose of ranitidine (300 mg) plus high nitrite/NDMA meals
  Ranitidine: Ranitidine 300 mg
  High nitrite/NDMA meals: Meals containing higher levels of nitrites and NDMA (cured meats diet)
- Placebo and Cured Meats Diet: Single dose of placebo plus high nitrite/NDMA meals
  Placebo: Oral placebo tablet
  High nitrite/NDMA meals: Meals containing higher levels of nitrites and NDMA (cured meats diet)
Arm/Group | Lead-in (No Treatment) | Ranitidine and Noncured Meats Diet | Placebo and Noncured Meats Diet | Ranitidine and Cured Meats Diet | Placebo and Cured Meats Diet
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/18 | 3/18 | 1/18 | 1/17 | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in (No Treatment) (N=18) | Ranitidine and Noncured Meats Diet (N=18) | Placebo and Noncured Meats Diet (N=18) | Ranitidine and Cured Meats Diet (N=17) | Placebo and Cured Meats Diet (N=17)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal gardnerella (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel Puncture Site Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT04397445/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04397445/SAP_001.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT04397445/ICF_002.pdf